CLINICAL TRIAL: NCT04309435
Title: DEcision-making Capacity: Intervention Development & Evaluation in Schizophrenia-spectrum Disorder: The DEC:IDES Trial
Brief Title: DEcision-making Capacity: Intervention Development & Evaluation in Schizophrenia-spectrum Disorder
Acronym: DEC:IDES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Edinburgh Napier University (Other)
Collaborators: King's College London (Other); University of Edinburgh (Other); University of Manchester (Other); Pennine Care NHS Foundation Trust (Other Government); Lancashire Care NHS Foundation Trust (Network); NHS Lothian (Other Government)
Responsible Party: Principal Investigator, Dr Paul Hutton, Associate Professor, Edinburgh Napier University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 1206004; HIPS/18/60 (Other Grant/Funding Number: Chief Scientist Office); 19/SS/0069 (Other: Scotland A Research Ethics Committee); 19/WA/0155 (Other: Wales Research Ethics Committee 5)
Record Dates: First submitted 2020-03-02; First posted 2020-03-16 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Schizophrenia and Related Disorders; Mental Competency
Keywords: schizophrenia; psychosis; umbrella trial; decision-making capacity; self-esteem; self-stigma; jumping to conclusions
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: This study is a pilot/feasibility Umbrella trial, comprising of 3 'interventionist-causal' trials (IC-RCTs).
Who Masked: Outcomes Assessor
Masking Description: Clinical research data will be gathered at baseline, post-intervention (week 8) and variable follow-up [week 24; only those randomised in the first 5 (England) to 8 (Scotland) months] by research assistants (RAs). RAs will be masked to group allocation to demonstrate to future funders this is achievable in an Umbrella trial. Blind-breaks will be recorded, and minimised using previously successful strategies (e.g., separate offices / diaries).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Self-esteem intervention (Experimental): The self-esteem intervention involves 6 x 1-hour therapy sessions, each of which will be provided by a fully trained and supervised psychological therapist over an 8-week period (to allow for cancelled appointments etc). It will involve the following elements:
  * Engagement and listening
  * Positive regard and empathy
  * Collaboration
  * Development of a shared understanding of low self-esteem (a 'psychological formulation')
  * Provision of written or audio-visual information relating to low self-esteem
  * Between-session activity for participant
  * Provision of structured self-help material relating to low self-esteem
  * Testing of beliefs related to low self-esteem
  * Practicing new strategies related to low self-esteem
  * Development of a shared plan to maintain gains in self-esteem
  Interventions: Behavioral: Self-esteem intervention
- Self-esteem control group (Placebo Comparator): 'Assessment and support' for participants with low self-esteem will also involve 6 x 1-hour sessions with a psychological therapist, over a period of 8 weeks. However, in these meetings, the therapist will work in collaboration with the person to complete a more detailed assessment of factors which help or hinder their decision-making capacity. They will provide engagement, listening, positive regard and empathy, but they will not develop a psychological formulation, nor will they provide the person with information relating to their problems. They will also not provide self-help material, or encourage the person to test their beliefs, practice new strategies or develop a shared plan for the future. Once the trial is over, however, the therapist will offer to meet with the person to share the results of the assessment and develop a psychological formulation. With the participant's consent, this information will also be shared with the clinical team.
  Interventions: Behavioral: Control procedure (assessment only)
- Self-stigma intervention (Experimental): The self-stigma intervention involves 6 x 1-hour therapy sessions, each of which will be provided by a fully trained and supervised psychological therapist over an 8-week period (to allow for cancelled appointments etc). It will involve the following elements:
  * Engagement and listening
  * Positive regard and empathy
  * Collaboration
  * Development of a shared understanding of high self-stigma (a 'psychological formulation')
  * Provision of written or audio-visual information relating to self-stigma
  * Between-session activity for participant
  * Provision of structured self-help material relating to self-stigma
  * Testing of beliefs related to self-stigma
  * Practicing new strategies related to self-stigma
  * Development of a shared plan to maintain reductions in self-stigma
  Interventions: Behavioral: Self-stigma intervention
- Self-stigma control group (Placebo Comparator): 'Assessment and support' for participants with high self-stigma will also involve 6 x 1-hour sessions with a psychological therapist, over a period of 8 weeks. However, in these meetings, the therapist will work in collaboration with the person to complete a more detailed assessment of factors which help or hinder their decision-making capacity. They will provide engagement, listening, positive regard and empathy, but they will not develop a psychological formulation, nor will they provide the person with information relating to their problems. They will also not provide self-help material, or encourage the person to test their beliefs, practice new strategies or develop a shared plan for the future. Once the trial is over, however, the therapist will offer to meet with the person to share the results of the assessment and develop a psychological formulation. With the participant's consent, this information will also be shared with the clinical team.
  Interventions: Behavioral: Control procedure (assessment only)
- Jumping to conclusions intervention group (Experimental): The 'jumping-to conclusions' (JTC) intervention involves 6 x 1-hour therapy sessions, each of which will be provided by a fully trained and supervised psychological therapist over an 8-week period (to allow for cancelled appointments etc). It will involve the following elements:
  * Engagement and listening
  * Positive regard and empathy
  * Collaboration
  * Development of a shared understanding of role of JTC (a 'psychological formulation')
  * Provision of written or audio-visual information relating to JTC
  * Between-session activity for participant
  * Provision of structured self-help material relating to JTC
  * Testing of beliefs related to JTC
  * Practicing new strategies related to reducing JTC
  * Development of a shared plan to maintain reductions in JTC
  Interventions: Behavioral: Jumping to conclusions intervention
- Jumping to conclusions control group (Placebo Comparator): 'Assessment and support' for participants who demonstrate the JTC bias will also involve 6 x 1-hour sessions with a psychological therapist, over a period of 8 weeks. However, in these meetings, the therapist will work in collaboration with the person to complete a more detailed assessment of factors which help or hinder their decision-making capacity. They will provide engagement, listening, positive regard and empathy, but they will not develop a psychological formulation, nor will they provide the person with information relating to their problems. They will also not provide self-help material, or encourage the person to test their beliefs, practice new strategies or develop a shared plan for the future. Once the trial is over, however, the therapist will offer to meet with the person to share the results of the assessment and develop a psychological formulation. With the participant's consent, this information will also be shared with the clinical team.
  Interventions: Behavioral: Control procedure (assessment only)

INTERVENTIONS:
Behavioral: Self-esteem intervention — See relevant study arm for description
  Arms: Self-esteem intervention
Behavioral: Self-stigma intervention — See relevant study arm for description
  Arms: Self-stigma intervention
Behavioral: Jumping to conclusions intervention — See relevant study arm for description
  Arms: Jumping to conclusions intervention group
Behavioral: Control procedure (assessment only) — See relevant study arms for description
  Arms: Jumping to conclusions control group; Self-esteem control group; Self-stigma control group

SUMMARY:
Treatment decision-making capacity ('capacity') refers to a person's ability to make decisions about their treatment. It is an important issue for people diagnosed with a schizophrenia-spectrum disorder ('psychosis') because impaired capacity can mean a person does not understand what treatment options are available, or the implications of those options.

In 2018 the National Institute of Health & Care Excellence (NICE) called for clinical trials of interventions such as talking therapies to help people regain capacity. However, running these trials can take several years. One way of reducing this delay is to run several trials at the same time, as part of one bigger trial called an 'Umbrella' trial. Although Umbrella trials have been used to accelerate the development of physical health interventions, they have yet to be used in mental health.

The main aims of this study are therefore to find out whether people with non-affective psychosis (schizophrenia-spectrum disorder) will take part in a single (rater) blind Umbrella trial of talking therapies to improve their treatment decision-making capacity (the DEC:IDES trial), and to understand their experiences of participation.

Before a larger version of the DEC:IDES trial can begin, it needs to be established that people with psychosis will want to take part in it. Specifically, the aim of this study is to establish whether they will stay in the trial until it is finished, or whether they will leave early. It will also examine why people might leave DEC:IDES early, so that it can be improved. For these reasons, a smaller version must be completed first. This will involve 3 small clinical trials, each with N=20 (Treatment N=10; Control N=10), each testing 1 of 3 different interventions. Each intervention has been designed to help participants resolve a problem which previous evidence suggests may reduce their decision-making ability. One intervention is designed to improve self-esteem, another is designed to reduce negative beliefs about psychosis ('self-stigma') and another is designed to help people with psychosis gather more information before making decisions.

The investigators will record how many people participate in and complete the trial, and they will ask people for their views on what they liked and did not like about taking part. All this information will help ensure the larger DEC:IDES trial is more acceptable to people with psychosis.

DETAILED DESCRIPTION:
1. BACKGROUND & RATIONALE FOR STUDY

   'Treatment decision-making capacity' ('capacity'), is defined as the ability to understand, appreciate, and retain information relating to a proposed treatment, weigh that information and communicate a choice. Capacity is now a pivotal concept in healthcare and law, and clinicians are legally obliged to respect patient autonomy where capacity exists.

   Capacity has been referred to as the 'gatekeeper of autonomy'. When it is lost there is a legal and ethical imperative for clinicians to work to support its return and retention. However in their scrutiny of capacity-law implementation, the United Kingdom (UK) House of Lords concluded: "Our evidence suggests that (supported decision-making) is rare in practice" and The United Nations Committee on the Convention on the Rights of Persons with Disabilities (UNCRPD) advised that greater provision of supported decision-making is essential if the UK is to be compliant with Article 12 of the Convention on Human Rights.

   Despite the importance and legal obligation to support capacity there is a lack of evidence on how to do this effectively. A recent systematic review and meta-analysis synthesised evidence from 23 studies on capacity in psychosis and found there were no randomised controlled trials (RCTs) of supported decision-making interventions. Psychiatrists view the evidence in this area as weak, and the National Institute for Health and Clinical Excellence (NICE) have called for RCTs to enhance evidence in this area. Anticipating this, over the last 5 years the research team, comprising clinicians, legal experts and researchers, have produced 5 systematic reviews and meta-analyses addressing various aspects of decision-making capacity in psychosis, and 5 clinical studies. These indicate that a lack of capacity is likely to stem from interactions between cognitive, emotional and social factors, the effects of which are moderated by a person's awareness of them. This model specifically predicts that 'self-stigma', low self-esteem, and the 'jumping to conclusions' (JTC) bias are likely to have large, additive adverse effects on their capacity.

   Psychological interventions that selectively reduce each of these hypothesised 'causal mechanisms' have already been developed. The next stage of this research is therefore to conduct 'interventionist-causal RCTs' (IC-RCTs) to examine whether these interventions can also cause improvements in capacity. Recommended to accelerate the development of treatments for psychotic symptoms such as delusions, these sophisticated trials are capable of producing invaluable information on what causes and improves impaired capacity. If the trials are run consecutively, people with psychosis could wait 10-15 years for definitive findings and would involve setting up several costly trial infrastructures to support each trial.

   One simple solution is to conduct these IC-RCTs concurrently, within one trial infrastructure. This approach, also known as an 'Umbrella trial', could produce results in half the time, for half the cost, meaning an effective capacity-supporting intervention could be produced in 5-6 years, rather than 10-15. The aim of this study is therefore to conduct the first Umbrella trial in mental healthcare, using this to accelerate the development of an intervention to support capacity in psychosis. However, prior to conducting a definitive trial, a variety of feasibility issues need to be examined in a randomised pilot study. The planned study addresses these.
2. AIMS & OBJECTIVES

   2.1. Aims & Linked Research Questions (RQs)

   Aim 1: Test data quality for a definitive trial (primary aim) (RQs 1,2,5); Aim 2: Test recruitment and retention rates for a definitive trial (RQs 2,3); Aim 3: Test trial procedures for a definitive trial (RQs 3,4); Aim 4: Assess acceptability of interventions for this group (RQs 3,4); Aim 5: Refine treatment protocols to ensure feasibility in clinical settings (RQs 3,4); Aim 6: Consolidate research infrastructure to support main trial (RQs 3,4).

   2.2. Research questions (RQs)

   RQ 1: What data quality and completion rates can be obtained for the main outcome measures? RQ 2: What proportion of eligible patients consent, engage, & complete the trial? RQ 3: What do participants, clinicians & collaborators think will improve study processes, including interventions? RQ 4: Are trial procedures acceptable to them, and feasible to implement? RQ 5: What sample size is required in a full study?
3. DESIGN & PROCEDURE

   3.1. Overview

   This study has been designed to find out whether participants can be recruited and retained in a larger trial characterised by the same design parameters (e.g., allocation ratio, blind assessment, types of treatment and control offered, multiple sites). The planned randomised pilot study is therefore a 20-month feasibility/pilot of a multi-site single (rater) blind Umbrella trial of psychological interventions to support treatment decision-making capacity in people diagnosed with non-affective psychosis (schizophrenia-spectrum disorders). It has been designed primarily to examine post-treatment (8 week) data retention rates for the planned primary outcome [MacArthur Competence Assessment Tool for Treatment (MacCAT-T) capacity ratings] in a future definitive trial. In this and the future study, participants will be randomly allocated to receive treatment as usual (TAU) plus a psychological intervention to improve either (i) self-stigma, (ii) self-esteem, or (iii) the jumping to conclusions reasoning bias, or TAU plus an attention control condition. RQs 3 & 4 will be addressed through qualitative interviews with participants and referrers/clinicians, using Framework analysis.

   Qualitative analysis of change in participant appreciation, as measured by the MacCAT-T, will be performed using qualitative case study methodology. MaCAT-T appreciation ratings will also be compared to ratings on the Expanded Schedule for the Assessment of Insight (SAI-E). Concordance between overall MacCAT-T judgements and pre and post clinical judgements of referring clinicians, assessed using a version of the Clinical Global Impression Scale (modified to assess global capacity ratings), will also be assessed.

   To minimise piloting costs 75% of the 60 patient participants will be recruited in the lead site (NHS Lothian). Each intervention group will be compared to its own control group (each receive the same standardised procedure) to ensure participants in each trial are equivalent with respect to their presenting mechanism.

   3.2. Participants & setting

   Adults (aged 18-65) diagnosed with schizophrenia-spectrum disorder with impaired treatment decision-making capacity, and presence of either low self-esteem, high self-stigma or the JTC bias will be recruited from inpatient and outpatient NHS mental health services across three UK sites; 75% from NHS Lothian; 12.5% from Pennine Care; 12.5% from Lancashire Care. Of these patient participants, 6 will be invited to attend a qualitative interview to understand their experiences of participating in the trial, as part of the Framework analysis. Up to a further 10 will be invited to attend a qualitative interview to understand and verify any change in their 'appreciation' of their illness and its treatment. Six clinical or social care staff who have either referred a participant to the study or have provided substantial care and treatment to a participant during the study, will also be invited to attend a qualitative interview to understand their experiences of the trial, again as part of the Framework analysis.

   3.3. Allocation, randomisation and assessment

   Allocation & randomisation: Participants will be assigned to one of the two-arm IC-RCTs based on whether they have predominantly low self-esteem (defined as scoring 14 or less on the Rosenberg Self-Esteem Inventory), high self-stigma (defined as scoring 60 or more on the Internalised Stigma of Mental Illness Scale), or the JTC bias (defined as selecting 2 or fewer beads on The Beads Task). Participants with multiple mechanisms will be randomly assigned. All participants will then be randomised (1:1) at the start of treatment session 1 to treatment or control, using randomised-permuted blocks of random size (block sizes of two or four), administered via a study-specific web-based portal according to a concealed randomisation sequence.

   Assessments: All participants will receive a full research assessment, by a Research Assistant (RA) masked to treatment group allocation, at week 0 (baseline) and week 8 (end of treatment). In addition to measures of change (see outcomes), the Clinical Interview for Psychotic Disorders and the Brief Neurocognitive Assessment will be administered to confirm diagnosis and assess cognitive functioning, respectively, at week 0. Participants randomised in the first 8 (Scotland) or 5 (England) months will be invited to complete a follow-up assessment at week 24. All qualitative interviews will be conducted with participants and their referrers/clinicians following the patient participants' 24-week assessment.

   3.4. Study interventions

   Active interventions (each 6 sessions over 8 weeks): Each intervention is structurally equivalent and will be delivered by the same therapist. The self-esteem intervention is informed by a previous protocol tested with people with persecutory delusions. The JTC intervention, developed and trialled by the researchers and colleagues previously, has been lengthened to 6 sessions by addressing positive beliefs about JTC decision-making and providing greater practice of non-JTC decision-making. The self-stigma intervention developed by a team including the current PI, has been reduced from 12 to 6 sessions by removing self-esteem focused elements.

   Inactive attention control (6 sessions over 8 weeks): The therapeutically inactive assessment component of a protocol developed and piloted previously by the researchers will be used. To maximise clinical benefit of participation, the potentially active component of this protocol (psychological formulation) will be provided, but only after the participant exits the trial.

   3.5. Data Analysis

   Quantitative: An independent statistician will conduct blind analysis of outcome data. Proportions, means, standard deviations, effect sizes and 95% confidence intervals for all time points will be reported descriptively, on both a strict intention-to-treat and per-protocol basis (≥50% attendance in treatment or control). Concordance between (a) MacCAT-T ratings and clinician ratings of capacity and (b) MacCAT-T appreciation ratings and SAI-E scores will be analysed.

   Qualitative: A trained RA will prepare topic guides, conduct, record and transcribe the interviews. Under supervision, the RA will also analyse the qualitative data following established guidelines for Framework analysis and qualitative case study methodology. For the Framework analysis, interviews with participants and referrers/clinicians will address feasibility and acceptability of the trial procedures, problems indicated in the quantitative data, and potential solutions. This ensures that the issue is not explored through one lens, but rather various lenses facilitating understanding about multiple facets of the phenomenon. For the qualitative case study analysis, interviews with participants will address their views on their diagnosis and treatment, any subjective change, and the participant's views on the reason for this change.

   3.6. Progression criteria for a full trial

   Funding for a larger trial, using the same trial design, will be sought if the target recruitment is met and post-intervention (8 week) MacCAT-T data from ≥75% of those randomised is retained. If this target is not met, findings from the Framework Analysis will be used to modify the design before further piloting and/or progression.

   3.7. Research Team & Expert Advisory Group

   This project will receive strong support from: (i) An Expert Advisory group, comprising of experts by experience, experts in law and policy, and experts in psychosis research; (ii) Professor Richard Emsley (Co-Investigator) is Professor of Trial Methodology and former Director of the Manchester Clinical Trials Unit. He sits on the Expert Advisory Group for the world-leading STAMPEDE Umbrella trial of interventions for prostate cancer; and (iii) An experienced multi-disciplinary research team selected to ensure experience and expertise in relation to the interventions, population, outcomes, methodology and ability to manage the various sites, and to strengthen their trial infrastructure for the later trial, building on their existing robust collaborations.
4. STUDY POPULATION

   4.1. Number of Participants and Sample Size Calculation

   The National Institute for Health Research (NIHR) guidance was used to calculate that 60 participants (average of 3-4 per month over 12-months) will allow for an estimated drop-out rate (i.e., data non-retention) of 15%, at week 8, to within a 95% confidence interval of +/- 9%. The proportion of people with schizophrenia-spectrum disorders and impaired capacity who have at least one of the proposed causal mechanisms is estimated to range from 80-100%. Pilot trials suggest ≥80% of those who have one of these mechanisms will consent and be randomised, ≥85% of whom will complete the trial. Six of the 60 participants and six of their referrers or clinicians will be invited to participate in a qualitative interview for the Framework analysis. Up to a further 10 of the 60 participants will be invited to participate in the qualitative interview for the qualitative case study of change in appreciation.

   4.2. Identification and Recruitment of Participants

   One pathway in which participants will be identified is through self-referral. To facilitate this, a poster will be placed in NHS mental health services to advertise the study. A study website will be available, including participant information sheets. Contact details will be provided for those interested in self-referral. Individuals who self-refer, will only be included in the study if they agree that a mental health professional involved in their care, can be contacted to obtain information for risk assessment purposes and to ensure participation is not contraindicated in some way. Another pathway in which participants will be identified is through clinician-referral. As per previous trials, local site Principal Investigators will support RAs to visit clinical services to present the trial, determine initial interest, and distribute information sheets. The information sheet will detail what participants are asked to do, how their information will be used and the possible risks and benefits of taking part in the study.

   For potential participants entering the study through self-referral, the RA will obtain their explicit verbal consent to contact their key worker/ care-coordinator to determine whether they meet inclusion criteria for the study and to conduct an initial risk assessment. The RA will also ask the clinical care team if they have any concerns about the potential participant's capacity to consent to take part in research. Should participants meet inclusion criteria for the study and continue to express an interest in taking part, the RA will contact them to arrange an appointment. All potential participants will have as long as they wish to consider the information sheet prior to being contacted by the RA, with a minimum period of 48 hours.

   For potential participants entering the study through the clinician-referral pathway, their clinicians will discuss the study with them and seek their verbal consent to pass their details on to the research team. A trained and supervised RA will then obtain contact details of potential participants from their clinicians and contact the potential participants directly to discuss the study further. Consenting participants will be given a participant information sheet and any initial questions will be answered. As in the self-referral case, consenting participants will be recontacted after a minimum period of 48 hours, with a longer period if required. They will also be risk assessed, and the eligible ones will participate in the trial.

   For those lacking research capacity, the same initial process will be followed. However in England, the opinion of the potential participant's Consultee will be sought, and in Scotland, consent from the appropriate person (see consent section) will be sought. In both countries, the study will not proceed if there is any indication that the potential participant objects to taking part.

   4.3. Consenting Participants

   During the first meeting with the potential participant, the RA will ensure they have received an information sheet. They will be given the option to review this again and answer any further questions. All potential participants will be reminded that participation is entirely voluntary and that deciding not to take part in the study will have no impact upon the clinical care they receive. They will also be informed of their right to withdraw from the study at any time, without giving a reason, and reassured that exercising their right to withdraw will have no impact upon the ongoing care they receive. Potential participants who still wish to take part will be asked to provide written informed consent at this stage. Once this has been completed, the study will commence. This process will be followed for referrers or clinicians who take part in the qualitative study but adapted to consider the fact that they are not receiving care or treatment. They will be assured that non-participation or withdrawal will have no effect on their employment.

   Capacity is decision-specific. This means capacity to consent to medication or a hospital admission is distinct from capacity to consent to research or psychological therapy. Nonetheless, a number of potential participants will lack the capacity to consent to both. As with a prior case-series, those with research capacity will be included, but specialist ethical approval to include those who lack it has also been secured.

   In Scotland, the legislative requirements of the Adults with Incapacity (Scotland) Act 2000, which makes provisions for research with this group will be followed. This means that in Scotland, Guardians, Welfare Attorneys or nearest relatives will be asked to provide consent on participants' behalf to taking part. They will be provided with Research Ethics Committee (REC) approved information sheets and consent forms. In England, the legislative requirements of the Mental Capacity (England and Wales) Act 2005, which also makes provisions for research with this group will be followed. This means that in England, Consultees will be asked to provide advice (which is binding on the researcher) as to whether a participant would wish to take part. They will be provided with a REC-approved information sheet and consultee declaration form.

   If a participant lacks capacity initially but regains it, their consent to continued participation in the study will be sought. Participants will be provided with a REC-approved continued participation information sheet and consent form designed for those who regain capacity. If a participant has capacity initially but loses it during the study, procedures for participants who lack capacity at the outset will be adhered to. This means that in Scotland, Guardians, Welfare Attorneys or nearest relatives will be asked to provide consent on participants' behalf so that they can continue participating in the study. Participants will be provided with a REC-approved continued participation information sheet and consent form. In England, Consultees will be asked to provide advice (which is binding on the researcher) as to whether a participant would wish to continue to take part. They will be provided with a REC-approved continued participation information sheet and consultee declaration form.

   A trained RA will, in conjunction with the Principal Investigator, determine whether participants have the capacity to give consent. The latter will ensure RAs and the Trial Manager attend NHS Scotland and NHS England training on informed consent and working with people who lack research capacity.

   4.4. Participant withdrawal

   Participants can withdraw from the study at any point, without giving any reason and without their legal rights or usual care being affected. Participants may also be withdrawn if their continuation is deemed to be harmful. The data monitoring and ethics committee (DMEC) will review all instances of adverse events, whether or not they are judged to be attributable to the trial or interventions, and, based on this information, determine whether the participant should be withdrawn. All events will be reported to the REC.

   Advance consent from all participants with capacity will be sought to retain existing data. This is in the event that they subsequently withdraw due to loss of contact, or loss of capacity to consent to research, where they have not otherwise informed the investigator that they wish their data to be removed. No data will be retained for individuals who lose capacity if the legal representative (Scotland) or Consultee (England) objects to this.
5. STUDY SUSPENSION OR DISCONTINUATION

   The research would be stopped in the event of a number of therapy-attributable adverse events. As earlier noted, any serious adverse events will be passed on to the independent DMEC for review and advice on whether to suspend or discontinue the study. This advice would be acted upon by the researchers, in consultation with the Sponsor and REC.
6. ADVERSE EVENTS

The interventions being tested have each been used previously with people with psychosis, including in randomised controlled trials and no severe adverse events have been reported. However, to improve the recording and reporting of adverse effects of psychological interventions, a robust protocol for assessing and managing any such risk will be completed at end of treatment and at follow-up by RAs masked to treatment condition.

This protocol, excluding the Adverse Events Questionnaire (which is designed to be completed after treatment), will also be completed by clinicians during the intervention (i.e., every session) to complete an assessment of severe adverse events. They will be instructed to report all adverse events to the trial manager, using a standardised form.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 18 and 65 years;
2. able to be interviewed and complete the measures;
3. diagnosed with a schizophrenia-spectrum disorder (schizophrenia, schizoaffective disorder, delusional disorder, psychosis not otherwise specified, brief psychotic disorder);
4. presumed or already judged to have impaired treatment decision-making capacity;
5. registered as patient with clinical or social care services

Exclusion Criteria:

1. have a moderate to severe learning disability;
2. have psychosis of a predominantly organic origin (e.g. brain injury, physical health condition, epilepsy) or have a primary diagnosis of substance or alcohol use disorder;
3. cannot understand English sufficiently to engage in conversation without an interpreter;
4. presents with a level of risk to others, including the researchers, that cannot be managed feasibility via suitable adjustments, as judged by Chief Investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-02-22 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited and randomised | Duration of recruitment window (12 months)
  This primary outcome relates to achieving the recruitment target (N=60). This will be defined as the overall number of participants recruited and randomised during the recruitment window, divided by the recruitment target.
MacArthur Competence Assessment Tool for Treatment (MacCAT-T) | Week 8 (end of treatment)
  This primary outcome refers to data completion rates at 8-weeks post-randomisation (end of treatment) on the MacCAT-T (anticipated primary outcome for a future trial). Data completion here refers to the number of participants completing MacCAT-T assessments at week 8 divided by the number of participants randomised. The MacCAT-T assesses participants on 4 domains:
  (i) Understanding scored 0-6 (3 items); (ii) Reasoning scored 0-8 (4 items); (iii) Appreciation scored 0-4 (2 items); and (iv) Expressing a choice scored 0-2 (1 items).
  Higher scores indicate greater current ability in each domain.

SECONDARY OUTCOMES:
MacArthur Competence Assessment Tool for Treatment (MacCAT-T) | Week 24 (variable follow-up)
  This outcome refers to data completion rates at 24-weeks post-randomisation (follow-up) on the MacCAT-T (anticipated primary outcome for a future trial). Data completion here refers to the number of participants completing MacCAT-T assessments at week 24 divided by the number of participants randomised AND eligible to receive a follow-up assessment [note: only those randomised in the first 5 (England) to 8 (Scotland) months] will be eligible for follow-up assessment]. The MacCAT-T assesses participants on 4 domains:
  (i) Understanding scored 0-6 (3 items); (ii) Reasoning scored 0-8 (4 items); (iii) Appreciation scored 0-4 (2 items); and (iv) Expressing a choice scored 0-2 (1 items).
  Higher scores indicate greater current ability in each domain.
Rosenberg Self Esteem Scale (RSE) | Weeks 0, 8 and 24 (variable follow-up)
  Retention and data completion rates on the Rosenberg Self Esteem Scale will be assessed. This scale has a minimum score of 0 and a maximum score of 30. Scores between 15-25 are considered normal, while scores <15 indicate low self esteem.
Semi-structured Interview Measure of Stigma (SIMS) | Weeks 0, 8 and 24 (variable follow-up)
  Retention and data completion rates on the Semi-structured Interview Measure of Stigma (SIMS) will be assessed. This interview measure has a minimum score of 0 and maximum score of 40, with higher scores indicating more severe self-stigma.
Beads task | Weeks 0, 8 and 24 (variable follow-up)
  Retention and data completion rates on the Beads Task will be assessed. Performance on the Beads Task is measured in 2 ways: (i) number of beads taken before a decision, and (ii) number of people making decisions based on 2 or fewer beads.
Number of deaths by suicide | Weeks 8 and 24 (variable follow-up)
  The number of deaths due to suicide occurring in each treatment and control group by week 8 and week 24 will be reported as part of the trial adverse event monitoring and reporting protocol.
Number of participants attempting suicide | Weeks 8 and 24 (variable follow-up)
  The number of participants attempting suicide and overall number of suicide attempts occurring in each treatment and control group by week 8 and week 24 will be reported as part of the trial adverse event monitoring and reporting protocol.
Number of participants experiencing suicidal crisis without suicide attempt | Weeks 0, 8 and 24 (variable follow-up)
  The number of participants experiencing suicidal crisis without attempting suicide and the overall number of suicidal crises occurring in each treatment and control group at weeks 0, 8 and week 24 will be reported as part of the trial adverse event monitoring and reporting protocol. Suicidal crisis without attempt is defined as a score of 2 on item 8 of the Calgary Depression Rating Scale for Schizophrenia (CDSS). Item 8 of the CDSS is scored 0 (absent) to 3 (severe), with higher scores indicating greater severity.
Calgary Depression Scale for Schizophrenia (CDSS) | Weeks 0, 8 and 24 (variable follow-up)
  Retention and data completion rates on the Calgary Depression Scale for Schizophrenia (CDSS) will be assessed. This 9-item interview measure has a minimum score of 0 and maximum score of 27, with higher scores indicating more severe depression.
Beck Anxiety Inventory (BAI) | Weeks 0, 8 and 24 (variable follow-up)
  Retention and data completion rates on the Beck Anxiety Inventory (BAI) will be assessed. This 21-item questionnaire measure has a minimum score of 0 and maximum score of 63, with higher scores indicating more severe anxiety.
Number of deaths not related to suicide | Weeks 8 and 24 (variable follow-up)
  The number of deaths not related to suicide occurring in each treatment and control group by weeks 8 and week 24 will be reported as part of the trial adverse event monitoring and reporting protocol.
Number of participants experiencing severe symptom exacerbation | Weeks 8 and 24 (variable follow-up)
  The number of participants experiencing severe symptom exacerbation at weeks 8 and 24 will be reported as part of the trial adverse event monitoring and reporting protocol. Severe symptom exacerbation is defined as a rating of ≥6 on the patient or researcher-rated Clinical Global Impression (CGI) and Clinical Global Impression Improvement (CGI-I) scales. Both the patient and researcher-rated CGI are scored from 1 to 7, with higher scores indicating greater symptom severity. Both the patient and researcher-rated CGI-I scales are scored from 1 to 7, with higher scores indicating less improvement.
Adverse Experiences in Psychotherapy (AEP) | Weeks 8 and 24 (variable follow-up)
  The Adverse Experiences in Psychotherapy (AEP) is a 28-item self-report measure that asks respondents to rate their agreement with statements regarding a variety of potential adverse events from participation in a psychotherapy trial (e.g., 'Taking part has made me feel more anxious'). Each statement is scored 0-4, with higher scores indicating greater agreement. For each statement, we will report the number of participants per group who rate provide a rating of 3 or 4 (corresponding to 'quite a lot' or 'very much'), at weeks 8 and 24.
Schizophrenia Quality of Life Scale (SQoLS) | Weeks 0, 8 and 24 (variable follow-up)
  Retention and data completion rates on the Schizophrenia Quality of Life Scale will be assessed. The scale consists of 30 items on 3 sub-scales:
  (i) Psychosocial (15 items); (ii) Motivation and energy (7 items); and (iii) Symptoms and side effects (8 items).
  Scores are transformed per scale to have a range from 0-100, higher scores indicating more significant difficulty/ poorer quality of life.
Questionnaire about the Process of Recovery (QPR) | Weeks 0, 8 and 24 (variable follow-up)
  Retention and data completion rates on the Questionnaire about the Process of Recovery will be assessed. The scale consists of 15 items and scores range from 0-30. Higher scores are indicative of recovery.
Brief Core Schema Scale (BCSS) | Weeks 0, 8 and 24 (variable follow-up)
  Retention and data completion rates on the Brief Core Schema Scale will be assessed.There are four scales. Participants first indicate whether they hold this belief (yes/no). If yes, they indicate on a scale from 1-4 how strongly they believe this. Higher scores indicate more strongly held beliefs.
  (i) negative beliefs about the self, (6 items), scored 0-24; (ii) negative beliefs about others, (6 items), scored 0-24; (iii) positive beliefs about the self, (6 items), scored 0-24; and (iv) positive beliefs about other, (6 items), scored 0-24.
Positive and Negative Syndrome Scale (PANSS) | Weeks 0, 8 and 24 (variable follow-up)
  Retention and data completion rates on the Positive and Negative Syndrome Scale will be assessed. The subscales of this interview measure are:
  (i) Positive symptoms (6 items) scored 6-42 (ii) Negative symptoms (8 items) scored 8-56 (iii) Excitement (4 items) scored 4-28 (iv) Emotional distress (5 items) scored 5-35 (v) Disorganised (7 items) scored 7-49
  Total score (30 items) ranges from 30-210. An adjusted scoring system (0-180) will be used in the current trial and numbers in each treatment and control group experiencing 0, 25%, 50%, 75% and 100% improvement will be calculated and reported in addition to means and standard deviations. Higher scores indicate more severe symptomatology on all scales.
Client Service Receipt Inventory (CSRI) | Weeks 0, 8 and 24 (variable follow-up)
  Retention and data completion rates on measures of service use will be assessed and reported using the Client Service Receipt Inventory. Each section is scored differently. Sections include information on number of inpatient days, number of contacts with outpatient services, medication & dose, criminal justice contacts, type and frequency of engagement with primary & community care contacts.
Number of blind-breaks | Weeks 0, 8 and 24 (variable follow-up)
  All blind-breaks will be recorded and reported to investigate feasibility of rater masking.

OTHER OUTCOMES:
Assessment of clinical validity of the MacArthur Competence Assessment Tool for Treatment (MacCAT-T) appreciation sub-scale | Duration of project (20 months)
  Up to 10 participants with improved MacCAT-T Appreciation subscale scores will be interviewed using qualitative 'case study' methodology to investigate the clinical validity of this change. MacCAT-T Appreciation ratings will be compared to ratings on the Expanded Schedule for the Assessment of Insight (SAI-E).The MacCAT-T Appreciation subscale is scored 0-4 (2 items), with higher scores indicating better appreciation. The SAI-E is scored from 0 to 14, with higher scores consistent with reduced insight, as defined by the SAI-E.
Assessment of clinical validity of the MacArthur Competence Assessment Tool for Treatment (MacCAT-T) overall judgements of capacity | Duration of project (20 months)
  Participants' clinicians will be asked to complete a version of the Clinical Global Impression Scale (CGI-capacity) at weeks 0 and 8, modified to assess treatment decision-making capacity. Concordance between CGI-capacity and MacCAT-T judgements of capacity will be assessed.The CGI-capacity is scored from 1 to 7, with higher scores indicating more severe decision-making incapacity. The MacCAT-T assesses participants on 4 domains:
  (i) Understanding scored 0-6 (3 items); (ii) Reasoning scored 0-8 (4 items); (iii) Appreciation scored 0-4 (2 items); and (iv) Expressing a choice scored 0-2 (1 items).
  Higher scores indicate greater current ability in each domain.
Participant, collaborator & clinical staff experience of trial | Duration of project (20 months)
  Using Framework Analysis, participants, collaborator and clinical staff experiences will be assessed and analysed vis-a-vis trial & intervention acceptability, including any suggested changes. Framework analysis is a qualitative methodology which facilitates the identification of converging and diverging information that arise from interview data, highlighting relationships between different parts of the data. It will be used to derive descriptive and/or explanatory conclusions around themes.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hutton, ClinPsyD, Study Director — Edinburgh Napier University
Locations (3):
- United Kingdom (3):
  - Pennine Care NHS Foundation Trust, Ashton-under-Lyne, Greater Manchester
  - Lancashire and South Cumbria NHS Foundation Trust, Preston, Lancashire
  - NHS Lothian, Edinburgh, Lothian

IPD SHARING:
Plan to Share IPD: No
Due to the small sample sizes involved, we will not share individual participant data with other researchers.

REFERENCES:
- [Derived] Hutton P, Taylor CDJ, Kelly J, Emsley R, Vikram A, Alexander CH, McCann A, Saddington D, Eliasson E, Burke J, Harper S, Karatzias T, Taylor PJ, Watson A, Dougall N, Stavert J, O'Rourke S, Glasgow A, Murphy R, Palmer K, Zaidi N, Bidwell P, Pritchard J, Carr L, Woodrow A. Accelerating the development of a psychological intervention to restore treatment decision-making capacity in patients with schizophrenia-spectrum disorder: An umbrella trial. Schizophr Res. 2025 Aug;282:184-197. doi: 10.1016/j.schres.2025.06.018. Epub 2025 Jul 3. PMID 40614350
- [Derived] Hutton P, Kelly J, Taylor CDJ, Williams B, Emsley R, Alexander CH, Vikram A, Saddington D, McCann A, Burke J, Eliasson E, Harper S, Karatzias T, Taylor PJ, Watson A, Dougall N, Stavert J, O'Rourke S, Glasgow A, Murphy R, Palmer K, Zaidi N, Bidwell P, Pritchard J, Carr L, Woodrow A. Accelerating the development of a psychological intervention to restore treatment decision-making capacity in patients with schizophrenia-spectrum disorder: a study protocol for a multi-site, assessor-blinded, pilot Umbrella trial (the DEC:IDES trial). Pilot Feasibility Stud. 2023 Jul 8;9(1):117. doi: 10.1186/s40814-023-01323-0. PMID 37422659
- See also: The DEC:IDES trial website — https://www.decides-trial.com/